CLINICAL TRIAL: NCT05602025
Title: An Open-Label, Randomized, Single-Dose, Multicenter, Parallel-Group Study to Compare the Pharmacokinetics of Subcutaneous Depemokimab When Delivered With a Safety Syringe Device or an Autoinjector in Healthy Adult Participants
Brief Title: A Study to Compare the Pharmacokinetics (PK) of Depemokimab When Delivered With a Safety Syringe Device (SSD) or an Autoinjector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214099
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: Autoinjector; Depemokimab; Healthy Participants; Safety Syringe Device; Pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a randomized, multicenter, open-label study in healthy adult participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving depemokimab via a SSD (Experimental)
  Interventions: Biological: Depemokimab
- Participants receiving depemokimab via an autoinjector (Experimental)
  Interventions: Biological: Depemokimab

INTERVENTIONS:
Biological: Depemokimab — Depemokimab will be administered via a SSD or autoinjector.

SUMMARY:
This study will compare the pharmacokinetics, safety, tolerability, and immunogenicity of Depemokimab administered via a SSD or autoinjector in healthy participants.

ELIGIBILITY:
Inclusion criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead electrocardiogram results.
* Body weight greater than or equal to (>=) 50 kilograms (kg) (110 pounds-mass/Ibs) and body mass index within the range 19 to 30 kg per meter square (inclusive).
* Women who have the potential to become pregnant must use a form of highly-effective contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study intervention, or interfering with the interpretation of data.
* Participants with allergy/intolerance to a monoclonal antibody or biologic or participants with a previous history of clinically significant multiple or severe drug allergies/intolerance.
* Current evidence or recent history of an infective illness.
* A positive pre-study drug/alcohol screen or a history (or suspected history) of alcohol misuse or substance abuse
* Clinically significant abnormalities.
* Positive test for severe acute respiratory syndrome coronavirus (SARS-CoV-2) at screening.
* Recent prior or concurrent clinical study experience.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of depemokimab | Up to Week 26
Area under the concentration-time curve from time zero extrapolated to infinity (AUC[0-inf]) of depemokimab | Up to Week 26

SECONDARY OUTCOMES:
Area under the concentration time curve from time zero to time of last observed quantifiable concentration (AUC[0-t]) of depemokimab | Up to week 26
Time to maximum observed plasma concentration (Tmax) of depemokimab | Up to Week 26
Apparent clearance following extravascular administration (CL/F) of depemokimab | Up to Week 26
Apparent volume of distribution following extravascular administration (Vd/F) of depemokimab | Up to week 26
Terminal elimination rate constant (lambda z) of depemokimab | Up to Week 26
Terminal elimination half life (T1/2) of depemokimab | Up to Week 26
Time of last measurable plasma concentrations (Tlast) of depemokimab | Up to week 26
Percentage of AUC(0-inf) due to extrapolation from Tlast to infinity (%AUCex) of depemokimab | Up to Week 26
Number of participants with presence of anti-drug antibody and neutralizing antibody to depemokimab | Pre-dose and Weeks 4, 8, 12, 26 post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/